CLINICAL TRIAL: NCT03470857
Title: Oxidative Stress and Inflammatory Processes in Selected Neoplasms in the Group of Oncological Patients Examined With the FDG PET/CT Method.
Brief Title: Oxidoreductive Balance and Lysosomal Activity in Cancer Patients.
Status: Completed | Type: Observational
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Paweł Sutkowy, Assistant professor, Nicolaus Copernicus University
Other Study IDs: KB 363/2017
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Neoplasms; Antioxidants; Oxidative Stress; Lipid Peroxidation; Inflammation; Lysosome Alteration
Keywords: Positron Emission Tomography Computed Tomography; Fluorodeoxyglucose F18; Cancer; Superooxide Dismutase; Catalase; Glutathione Peroxidase; Malondialdehyde; Conjugated Dienes; Acid Phosphatase; Cathepsin D; Alpha-1-Antitrypsin; Arylsulfatase; 8-iso-Prostaglandin F2alpha; 4-Hydroxynonenal; Total Antioxidant Capacity; Vitamin A; Vitamin E
MeSH Terms: conditions — Neoplasms; Inflammation; Ceroid Lipofuscinosis, Neuronal, 10; alpha 1-Antitrypsin Deficiency | interventions — Immunocompromised Host

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood collected from the basilic vein from the study participants into two vacuum test tubes only once (from patients during FDG PET-CT diagnosis): for full blood (K2EDTA) and blood serum (clot activator and gel separator).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Oncological patients: lymphomas (Hodgkin's, DLBCL), breast and ovarian cancers, brain gliomas.
  Interventions: Diagnostic Test: Patients
- Control: The number at most half as large as the patients' group, composed of healthy people at similar age and the same sex as patients.

INTERVENTIONS:
Diagnostic Test: Patients — The FDG PET/CT imaging will be performed as part of typical medical procedures related to the diagnosis and monitoring of cancers at the Oncology Center in Bydgoszcz, Poland
  Groups: Patients

SUMMARY:
The research aims to determine the parameters of oxidative stress and inflammatory processes and compare these parameters with the image obtained using positron emission tomography (PET) with 2-deoxy-2-[fluorine-18]fluoro- D-glucose (18F-FDG) integrated with computed tomography (CT) in the group of oncological patients.

DETAILED DESCRIPTION:
FDG PET/CT is very sensitive imaging tool for the detection of neoplasms. Neoplasm tissue is characterized by a much higher level of metabolism than healthy tissues, therefore a 95% cases of use the method regard oncology. Fluorodeoxyglucose (FDG) is absorbed by patients' organism as glucose but it does not undergo metabolism. The increased degree of FDG accumulation in tissue means its higher metabolic activity. FDG accumulates in the tumor tissue and radiates enabling its detection but the substance has not been shown to be harmful to patient at doses used in the diagnostics.

Tumor formation is a multi-stage process in which the phases of initiation, promotion and progression are distinguished. Neoplastic transformation of healthy cells is associated with disturbances of the cell cycle caused by mutations of proto-oncogenes (activation of cell division) and/or suppressor genes (blocking cell division) and mutator genes (protecting the DNA against damage or its repairing) under the influence of various factors. Increasing data indicate that one of the most important factors initiating neoplasm are reactive oxygen species (ROS) and oxidative stress. Mechanisms responsible for induction of oxidative stress in cancer cells are not fully explained. It is known that they are closely related to inflammation, as well as intense cellular metabolism associated with continuous proliferation, mutations in the genetic material and dysfunctions in the mitochondrial respiratory chain.

In this study a number of markers of oxidative stress and inflammation are planned to be determined including: the activities of antioxidant and lysosomal enzymes, as well as concentrations of lipid peroxidation products and low molecular weight antioxidants. The PET/CT imaging will be performed as part of standard medical procedures related to the diagnosis and monitoring of cancer diseases at the Oncology Center in Bydgoszcz, Poland.

ELIGIBILITY:
Inclusion Criteria:

- sign informed consent form for participation in the study

Exclusion Criteria:

* other diseases,
* bad feeling of the studied individual on the day of the study,
* the participants will not be minor and incapacitated persons, soldiers, prisoners and persons dependent in any way from the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Oncology Center in Bydgoszcz, Poland, who suffer from: lymphomas (Hodgkin's, DLBCL), breast and ovarian cancers and brain gliomas. The patients report to the Oncology Center for PET-CT diagnosis.
  Control group: similar age and the same sex as the patients; number: the half number of the patients.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Superoxide Dismutase | 1 day (Single measurement)
  Antioxidant enzyme
Catalase | 1 day (Single measurement)
  Antioxidant enzyme
Glutathione Peroxidase | 1 day (Single measurement)
  Antioxidant enzyme
Thiobarbituric acid reactive substances (Malondialdehyde) | 1 day (Single measurement)
  Secondary lipid peroxidation product
Conjugated Dienes | 1 day (Single measurement)
  Primary lipid peroxidation product
8-iso-Prostaglandin F2alpha | 1 day (Single measurement)
  Secondary lipid peroxidation product
4-Hydroxynonenal | 1 day (Single measurement)
  Secondary lipid peroxidation product
Total Antioxidant Capacity | 1 day (Single measurement)
  Total antioxidant potential of blood serum in the participant
Acid Phosphatase | 1 day (Single measurement)
  Lysosomal enzyme
Cathepsin D | 1 day (Single measurement)
  Lysosomal enzyme
Arylsulfatase | 1 day (Single measurement)
  Lysosomal enzyme
Alpha-1-Antitrypsin | 1 day (Single measurement)
  Serine protease inhibitor
Vitamins A and E | 1 day (Single measurement)
  Low molecular weight antioxidants

SECONDARY OUTCOMES:
FDG PET/CT scanning | 1 day (Single measurement)
  Positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose integrated with computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Sutkowy, PhD, Principal Investigator — The Chair of Medical Biology, Collegium Medicum of Nicolaus Copernicus University
Locations (3):
- Poland (3):
  - The Chair of Medical Biology, Collegium Medicum of Nicolaus Copernicus University, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Department of Nuclear Medicine of Center Oncology in Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Department of Positron Emission Tomography and Molecular Diagnostics, Collegium Medicum of Nicolaus Copernicus University, Bydgoszcz, Kuyavian-Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: No
There is no the individual participant data (IPD) sharing plan.